CLINICAL TRIAL: NCT01735006
Title: A Phase III Multicenter, Randomized, Double-Blind, Placebo(Hepatitis E Vaccine)Controlled Study to Evaluate the Efficacy, Immunogenicity and Safety of a Recombinant(E.Coli)Human Papillomavirus Bivalent Vaccine in Healthy Women
Brief Title: Efficacy and Immunogenicity Study of Recombinant Human Papillomavirus Bivalent（Type 16/18 ）Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry); Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Jun Zhang, professor, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV-PRO-003
Record Dates: First submitted 2012-11-18; First posted 2012-11-28 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Human Papillomavirus 16; Human Papillomavirus 18; vaccine; Cervical Intraepithelial Neoplasia; cervical Cancer; Vaginal intraepithelial neoplasia; Vulvar intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection | interventions — Papillomavirus Vaccines; hecolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV vaccine (Experimental): This dosage contains 40μg HPV 16 virus-like particle antigen and 20μg HPV 18 virus-like particle antigen adsorbed in alum-adjuvant
  Interventions: Biological: HPV Vaccine
- HEV vaccine (Placebo Comparator): commercialized HEV vaccine which contains 30μg HEV antigen adsorbed in alum-adjuvant
  Interventions: Biological: HEV vaccine

INTERVENTIONS:
Biological: HPV Vaccine — 3 doses at month 0,1 and 6
  Arms: HPV vaccine
Biological: HEV vaccine — 3 doses at month 0,1 and 6
  Other Names: Hecolin
  Arms: HEV vaccine

SUMMARY:
This is a Phase III clinical trial of the novel recombinant HPV 16/18 bivalent vaccine manufactured by Xiamen Innovax Biotech CO., LTD. The primary objective of this study is to demonstrate the efficacy of the vaccine against relevant outcomes in healthy women above 18 years old at enrolment. The secondary objectives are to evaluate the safety, immunogenicity and immuno-persistence of the vaccine. Meanwhile, this study tries to compare the difference of safety and immunogenicity among different lots. Approximately 6000 study subjects will be enrolled and randomly stratified into 2 groups and receive human papillomavirus (HPV) vaccine(three different lots) or commercialized hepatitis E vaccine(Hecolin) according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects between, and including, 18 and 45 years of age at the first vaccination;
2. Healthy subjects as established by medical history and history-oriented clinical examination;
3. Be able to understand and comply with the request of the protocol;
4. Without acute cervicitis;
5. Not pregnant;
6. Have intact cervix.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine)within 30 days preceding the first vaccination, or plan to use during the study period;
2. Are using immunosuppressants;
3. Administration of immunoglobulin and/or any blood products within the three months preceding the first vaccination or planned administration during the study period;
4. Vaccinated of inactivated vaccine 14 days or attenuated vaccine 21 days before the enrollment;
5. Fever;
6. Concurrently participating another clinical trial;
7. Has received vaccines against HPV 16/18 ;
8. Immunodeficient;
9. History of allergic disease;
10. Serious medical disorders;
11. Blood coagulation disorders;
12. Epilepsy;
13. Unable to comply with protocol due to the mental illness;
14. Visible Condyloma;
15. Pregnant or breast-feeding women;
16. vergins;
17. Have more than 4 sexual partners.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7372 (Actual)
Dates: Start 2012-11-22 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Histopathologically-confirmed CIN2+ and/or VIN2+ and/or VaIN2+ Associated With HPV-16 and/or -18 Cervical Infection | expected 5-6 years
Number of Subjects With HPV-16 and/or -18 persistent cervical infection(6-month+ definition) | expected 2-3 years

SECONDARY OUTCOMES:
Number of Subjects Reporting Solicited Local and General Symptoms | Within 7 days after each vaccination
Number of Subjects Reporting Unsolicited Adverse Events | Month 7
Number of Subjects Reporting Serious Adverse Events (SAEs) | expected 5-6 years
number of subjects with persistent cervical infection (12-month+ definition)associated with HPV-16 and/or HPV-18 | expected 5-6 years
number of subjects Histopathologically-confirmed CIN1+ and/or VIN1+ and/or VaIN1+ associated with HPV-16 and/or -18 cervical infection | expected 5-6 years
number of subjects with incidence infection associated with HPV-16 and/or HPV-18 | expected 2-3 years
Anti-HPV16 and anti-HPV18 seroconversion rates and geometric mean concentrations at Months 7 | month 7

OTHER OUTCOMES:
Number of subjects histopathologically confirmed CIN2+ and/or VIN2+ and/or VaIN2+ associated with oncogenic HPV types | expected 5-6 years
  Histopathologically confirmed CIN2+ and/or VIN2+ and/or VaIN2+ associated with oncogenic HPV types (e.g. HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68) detected within the lesional component of the tissue specimen (by PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Youlin Qiao, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Ting Wu, Ph. D, Study Director — Xiamen University
Locations (1):
- Cancer Institute ＆ Hospital Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Derived] Liao M, Quan J, Zhu K, Hu X, Shen S, Xu J, Nie C, Xu W, Jiang H, Wu X, Zhong Y, Peng Y, Cai S, Chen J, Zhang C, Lin B, Su Y, Huang S, Chen Q, Wu T, Zhang J, Xia N. Immunopersistence of one or two doses of an Escherichia coli produced bivalent HPV vaccine. NPJ Vaccines. 2025 Dec 17. doi: 10.1038/s41541-025-01335-2. Online ahead of print. PMID 41407728
- [Derived] Zhao FH, Wu T, Hu YM, Wei LH, Li MQ, Huang WJ, Chen W, Huang SJ, Pan QJ, Zhang X, Hong Y, Zhao C, Li Q, Chu K, Jiang YF, Li MZ, Tang J, Li CH, Guo DP, Ke LD, Wu X, Yao XM, Nie JH, Lin BZ, Zhao YQ, Guo M, Zhao J, Zheng FZ, Xu XQ, Su YY, Zhang QF, Sun G, Zhu FC, Li SW, Li YM, Pan HR, Zhang J, Qiao YL, Xia NS. Efficacy, safety, and immunogenicity of an Escherichia coli-produced Human Papillomavirus (16 and 18) L1 virus-like-particle vaccine: end-of-study analysis of a phase 3, double-blind, randomised, controlled trial. Lancet Infect Dis. 2022 Dec;22(12):1756-1768. doi: 10.1016/S1473-3099(22)00435-2. Epub 2022 Aug 26. PMID 36037823